CLINICAL TRIAL: NCT04871009
Title: A Trial of Neurofeedback as an Adjunctive Treatment for Youth in Outpatient Mental Health Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Thomas O'Connor, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00006013
Record Dates: First submitted 2021-04-28; First posted 2021-05-04 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-09

CONDITIONS: Trauma
MeSH Terms: conditions — Wounds and Injuries | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Placebo Comparator): routine clinical psychotherapy
  Interventions: Behavioral: standard of care
- Neurofeedback Intervention plus standard of care (Experimental): routine clinical psychotherapy plus 3 to 4 neurofeedback interventions per week.
  Interventions: Behavioral: Neurofeedback Intervention; Behavioral: standard of care

INTERVENTIONS:
Behavioral: Neurofeedback Intervention — InteraXon, Inc. produces the MUSE 2 wearable neurofeedback device and mobile application (heretofore referred to as the "MUSE app"), respectively comprising the electroencephalogram (EEG) hardware and interactive software components that will be used in this intervention. The MUSE 2 is an adjustable headband that is placed across the forehead and over and behind the ears. It contains EEG sensors for active sites across the forehead and behind the ears, and an additional reference site behind the ear. These sensors use EEG technology to passively record children's brainwaves. During a session, caregivers will help children place the MUSE 2 on their heads and connect it to the app on their personal device. Children's brain activity is recorded by the MUSE 2 and is represented on the app through audio-based feedback that children will listen to with earbuds, and use their volition to influence in real time, with the goal of gaining increased control over their own brain activity.
  Arms: Neurofeedback Intervention plus standard of care
Behavioral: standard of care — trauma focused cognitive behavioral therapy or other behavioral therapy at the discretion of therapist

SUMMARY:
The purpose of this study is to test the feasibility and effectiveness of a neurofeedback intervention conducted as an adjunctive behavioral health treatment to reduce trauma and affective symptoms in trauma-exposed youth.

ELIGIBILITY:
Inclusion Criteria:

(children)

* caregiver-reported exposure to two or more ACE types on the ACE-Q-Child measure.
* ages of 6-12 years old
* receiving or eligible to receive trauma-focused cognitive behavior therapy or another type of trauma-focused therapy, as determined by their primary therapist, designated as the TAU condition
* speaks and reads English

(caregivers)

* own an iPhone, iPad, smartphone, or tablet that is equipped with Bluetooth and uses an Apple or Android operating system that is compatible with the MUSE Calm app and accompanying MUSE wearable neurofeedback device
* speaks and read English

Exclusion Criteria:

Child-caregiver dyads will be excluded if

* the child falls outside of the required age range,
* has a documented history of epilepsy
* is currently considered to be at high risk for suicide attempt
* is currently experiencing psychosis

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Mean change in Trauma Symptom Checklist for Young Children (TSCYC) | baseline to 3 months
  Children's trauma symptoms will be measured by the Trauma Symptom Checklist for Young Children (TSCYC) at baseline and post-intervention intervals. This caregiver-report measure is developed for children between the ages of 4-12. It consists of 90-items that encompass two reporter validity scales, eight symptom-specific clinical subscales. Answers to individual items are based on a 4-point scale with response options ranging from 1 ("Not at All") to 4 ("Very Often"), and is administered and scored in accordance with manualized instructions. This study will assess trauma symptoms via subscale scores for levels of overall post-traumatic stress, dissociation, post-traumatic intrusion, arousal, and avoidance, and trauma-related aggression. Scale ranges from 90-360 with higher scores indicating worse outcomes.
Mean change in Short Mood and Feelings Questionnaire (SMFQ) | baseline to 3 months
  The child-report version of the Short Mood and Feelings Questionnaire (SMFQ)contains 13 items measuring depressive symptom severity over a 2-week period. Each item has 3 response categories: "True" (=2, the item applies to them most of the time), "Sometimes" (=1, the item applies to them sometimes), or "Not True" (=0, the item is not true about them). Scale ranges from 0-26 with higher scores indicating worse outcome.
Mean change in Patient Reported Outcomes Measurement Information System Pediatric Item Bank v2.0 - Anxiety - Short Form 8a (PROMIS) | baseline to 3 months
  The child-report version of the Patient Reported Outcomes Measurement Information System Pediatric Item Bank v2.0 - Anxiety - Short Form 8a (PROMIS)measures anxiety symptoms experienced by youth over the past seven days (PROMIS, 2019). The PROMIS (2019) contains 7 items, each with a 5-point Likert scale (1-5) by which youth indicate the frequency that each item applies to them (1=Never, 2=Almost Never, 3=Sometimes, 4=Often, 5=Almost Always). Scales ranges from 1-35 with higher scores indicating worse outcome.

SECONDARY OUTCOMES:
Number of caregivers reporting childhood trauma | baseline to 3 months
  Caregivers will be asked to respond yes or no to the same questions asked on the Center for Youth and Wellness Adverse Childhood Experiences (CYW ACE-Q) this time with respect to their own childhoods.
  This is a 17-item, yes/no, child-specific (ages 0-12) version of a measure that includes 10 items on abuse, neglect, and household dysfunction. These items comprise section 1 of the measure. Seven additional items comprise section 2 of the measure and include foster care placement, bullying, death of a primary caregiver, separation from primary caregiver due to deportation or immigration, serious medical procedure/illness, witnessing neighborhood violence, and experiencing discrimination. If any items are reported, the caregiver will be categorized as having reported trauma.
Mean number of sessions per week | 3 months
  A weekly check in survey will be used to collect the number of sessions per week and the duration of each session.
Mean satisfaction with the intervention | 3 months
  A weekly check in survey will be used for caregivers to rate their satisfaction with the intervention on a 5-point scale (1 = very dissatisfied; 5 = Very Satisfied). The scale ranges from 1-5 with 5 indicating higher satisfaction.
mean length of each session | 3 months
  A weekly check in survey will be used to collect from caregivers the number of sessions per week and the duration of each session.
Mean change in Beck Depression Inventory II (BDI-II) | baseline to 3 months
  Beck Depression Inventory II (BDI-II) that assesses symptoms of depression over the prior two-week period in accordance with DSM-IV diagnostic criteria for major depressive disorder. The BDI-II is acceptable for use with clinical and non-clinical populations. It contains 21 items, each with a four-point response scale ranging in severity from no symptoms (1) to severe symptoms (3). A cut-off score of 20 is used to indicate depression among non-clinical populations, while scores ranges of 0-13 (minimal depression), 14-19 (mild depression), 20-28 (moderate depression), and 29-63 are used to assess levels of depression among clinically diagnosed patients. The scale ranges from 0-63 with higher scores indicating worse outcomes.
post traumatic stress disorder (PTSD) Checklist for DSM-5 (PCL-5) | baseline to 3 months
  The post traumatic stress disorder (PTSD) Checklist for DSM-5 (PCL-5) is a validated screening instrument that measures past-month post traumatic stress disorder symptoms. The PCL-5 contains 20 items scored on a 5-point Likert scale, in which respondents indicate their agreement with each item, ranging from 0 ("Not at All") to 4 ("Extremely"). The scale ranges from 0-80 with higher scores indicating worse outcome.
Parental Stress Scale (PSS) | Baseline to 3 months
  The Parental Stress Scale (PSS) is an 18-item measure that assesses parenting-related stress among caregivers. Each item contains 5 numbered response options, ranging from 1 ("Disagree Strongly") to 5 (Strongly Agree), along with an additional "Not Sure" option. The scale ranges from 18-90 with higher scores indicating worse outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided